CLINICAL TRIAL: NCT05998668
Title: The Effect of Genital Hygiene Training Provided to Turkish Women Living in Rural Areas With a Vulvovaginal Candidiasis History on Genital Hygiene Behaviors and Self-care Agency
Brief Title: Genital Hygiene Training Provided to Turkish Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assistant professor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/3782
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Genital Hygiene; Genital Hygiene Behaviors; Self-care Agency
Keywords: genital hygiene; vulvovaginal candidiasis; genital infection; self-care; rural area
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Intervention Model Description: The study was desined as a randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- genital hygiene training (Experimental): Following the pretest, "genital hygiene behaviors training" was provided to the women in the intervention group by E.S.B., one the researchers. In addition, a genital hygiene brochure prepared by the researchers which included the same content as the training was given to each participant. The training program was carried out as oral instruction as well as using the demonstration method which is called as "tell-show-do". Individual questions of the women were answered at the end of the training. In the first meeting with the women, 2 sessions of 45 minutes with a 10-minute break were held in the counselling rooms of the relevant family health centers. Four weeks after these sessions, a 45-minute session was held in order to reinforce the training with the same method. Four weeks after the data collection tools used in the research were filled in as a pre-test, post-test data were obtained with the same measurement tools.
  Interventions: Other: Genital hygiene training
- Routine checks (No Intervention): The researchers applied no initiative to the control group, and the women in the control group solely had the routine checks. The women in the control group filled out all pretest forms (A sociodemographic questionnaire, Genital Hygiene Behavior Inventory (GHBI), and Self-Care Agency Scale (SCAS). The post-test forms (GHBI, SCAS) were re-administered 4 weeks later to women who did not receive any intervention.

INTERVENTIONS:
Other: Genital hygiene training — In the first meeting with the women, 2 sessions of 45 minutes with a 10-minute break were held in the counselling rooms of the relevant family health centers. Two weeks after these sessions, a 45-minute session was held in order to reinforce the training with the same method.
  Arms: genital hygiene training

SUMMARY:
Purpose: In the study, it was aimed to determine the effect of genital hygiene training provided to women living in rural areas with a vulvovaginal candidiasis history on genital hygiene behaviors and self-care agency.

Material and methods: This study with a randomized controlled design was conducted with the participation of women who were registered to Family Health Centers located in two villages in the rural areas in the east of Turkey and who had a history of vulvovaginal candidiasis within the last year. The study sample consisted of 114 women in total, 57 of whom were in the intervention group and 57 were in the control group. The women in the intervention group were provided with genital hygiene behaviors training. The study data were collected Identifying Information Form, Genital Hygiene Behavior Inventory (GHBI), and Self-Care Agency Scale (SCAS).

DETAILED DESCRIPTION:
Design The study was designed as a randomized controlled trial in which the subjects were randomly assigned to the intervention (receiving genital hygiene training) and the control group.

The study was conducted in the Family Health Centers of two randomly selected villages with a distance of 20-30 km to Van province located in the east of Turkey. These villages are in a rural area and people make their living mostly through farming. Each village had one family health center, and other health institutions were in the provincial center. Family health centers are primary care health institutions which provide reproductive health service for women (healthy woman follow-up, laboratory tests, family planning, education, counselling, etc.). While training is provided within the scope of preventive health services in family health centers, there is no training provided specifically on genital health regarding vulvovaginal candidiasis. Working hours are between 08.00-17.00 every weekday, and there are three family health doctors and three family health professionals (midwife and/or nurse) in these centers.

Sample The study sample consisted of women who tested positive on at least one culture test and received and completed treatment for vulvovaginal candidiasis in the last year according to the registry of the Family Health Centers. The study inclusion criteria were being within the age range of 18-49 years, not having a systemic disease, and not being pregnant or puerpera between the dates when the study was conducted. According to the registration system of the family health centers, 1,400 women who met these criteria were receiving service from these centers.

In order to predict the most suitable sample size for the study, priori-power analysis was performed on a web-based software (https://www.stat.ubc.ca/~rollin/stats/ssize/n2.html). Sample size was calculated to be 57 for each group (57 in the intervention group and 57 in the control group) with 5% margin of error at two-way significance level, 95% confidence interval, 80% power of representing the population and by assuming that the mean score of genital hygiene behaviors, which was 84.51 (standard deviation 5.69), would increase by three points. According to the records of the family health centers where the study was conducted, there were 142 women who received and completed treatment for vulvovaginal candidiasis in the last six months. 142 women were assigned to the intervention and control groups through randomization. Women were listed by the researchers for randomization. According to the list, women with odd numbers were assigned to the intervention group and those with even numbers were included in the control group. The sample selection process carried out in line with CONSORT criteria is presented in Figure 1.

Data Collection Tools In the collection of the study data, Identifying Information Form, Genital Hygiene Behavior Inventory (GHBI), and Self-Care Agency Scale (SCAS) were used.

Identifying Information Form: The form developed by reviewing the literature consisted of questions inquiring about the sociodemographic characteristics of the women (age, educational status, employment status, etc.).

Genital Hygiene Behavior Inventory (GHBI): The scale was developed in Turkish in order to measure genital hygiene behaviors of women, and the validity and reliability study of the scale was conducted by Karahan in 2017. The scale consists of three subscales, which are "general hygiene" (12 items), "menstrual hygiene" (8 items), and "abnormal finding awareness" (3 items). The 23-item and 5-point Likert type scale is scored between 1 and 5. The minimum and maximum scores to be obtained from the scale are 23 and 115. As the score obtained from the scale increases, the women's levels of displaying proper genital hygiene behaviors increase. The Cronbach's alpha internal consistency coefficient of the scale is 0.80.

Self-Care Agency Scale (SCAS): The scale was developed by Kearney and Fleischer in 1979. The Turkish validity and reliability of the scale was conducted by Nahcivan in 1993. It is used to measure individuals' self-care agency levels. Each item of the 35-item and 5-point Likert type scale is scored between 0 ad 4. The minimum and maximum scores to be obtained from the scale are 0 and 140. A high score on the scale shows the individual's high level of self-care agency. The Cronbach's alpha internal consistency of the scale is 0.89.

Procedures The women assigned to the intervention and control groups were called on their telephone numbers registered at the family health center by the researchers to inform them about the study, and they were invited to the family health centers. The pretest data were obtained from the women through the scales used in the study and the questionnaire on their sociodemographic characteristics by face-to-face interviews held by the researchers in the counselling room in the family health centers. Four weeks later, posttest data were collected by following the same procedures.

Following the pretest, "genital hygiene behaviors training" was provided to the women in the intervention group by E.S.B., one the researchers. In addition, a genital hygiene brochure prepared by the researchers which included the same content as the training was given to each participant. The training program was carried out as oral instruction as well as using the demonstration method which is called as "tell-show-do". Individual questions of the women were answered at the end of the training. In the first meeting with the women, 2 sessions of 45 minutes with a 10-minute break were held in the counselling rooms of the relevant family health centers. Two weeks after these sessions, a 45-minute session was held in order to reinforce the training with the same method. No intervention was made to the women in the control group.

Genital hygiene training program was developed by reviewing the literature, and expert opinion was taken for content check before application. In line with the opinions of three academics in the field of nursing, necessary corrections were made, and the training program was finalized. The training program included introduction of reproductive organs, properties of genital discharge, achieving hand and general hygiene, genital infections, hygiene rules in sexual contact, ensuring genital hygiene during menstruation, problems related to genital organs, and coping with genital problems.

ELIGIBILITY:
Inclusion Criteria:

* women who tested positive on at least one culture test and received and treatment for vulvovaginal candidiasis in the last year according to the registry of the Family Health Centers, within the age range of 18-49 years, not having a systemic disease, and not being pregnant or puerpera between the dates when the study was conducted.

Exclusion Criteria:

* Those who cannot communicate in Turkish, who are illiterate

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women between the ages of 18-49 years
Enrollment: 114 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Genital Hygiene Behavior Inventory (GHBI) | Change from genital hygiene behavior levels at 4 weeks
  The scale was developed in Turkish in order to measure genital hygiene behaviors of women, and the validity and reliability study of the scale was conducted by Karahan in 2017. The scale consists of three subscales, which are "general hygiene" (12 items), "menstrual hygiene" (8 items), and "abnormal finding awareness" (3 items). The 23-item and 5-point Likert type scale is scored between 1 and 5. The minimum and maximum scores to be obtained from the scale are 23 and 115. As the score obtained from the scale increases, the women's levels of displaying proper genital hygiene behaviors increase.

SECONDARY OUTCOMES:
Self-Care Agency Scale (SCAS) | Change from self-care agency levels at 4 weeks
  The scale was developed by Kearney and Fleischer in 1979. The Turkish validity and reliability of the scale was conducted by Nahcivan in 1993. It is used to measure individuals' self-care agency levels. Each item of the 35-item and 5-point Likert type scale is scored between 0 ad 4. The minimum and maximum scores to be obtained from the scale are 0 and 140. A high score on the scale shows the individual's high level of self-care agency.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Sabanci Baransel, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No